CLINICAL TRIAL: NCT00002835
Title: A Randomized Prospective Study of Early Intensification Versus Alternating Triple Therapy for Patients With Poor Prognosis Lymphoma
Brief Title: Combination Chemotherapy in Treating Patients With Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDA DM95-121; P30CA016672 (NIH); MDA-DM-95121 (Other: UT MD Anderson Cancer Center); NCI-V96-1010; CDR0000065044 (Registry Identifier: NCI PDQ); NCT00038740 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2003-04-16 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Lymphoma
Keywords: stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic | interventions — Bleomycin; Filgrastim; Granulocyte Colony-Stimulating Factor; Interferon-alpha; Carmustine; Cisplatin; Cyclophosphamide; Cytarabine; Etoposide; Idarubicin; Ifosfamide; Leucovorin; Melphalan; Methotrexate; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; Mitoxantrone; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): 3 courses of early intensification:
  First course: Ifosfamide (IFF) IV continuously and Etoposide (VP-16) IV over 2 hours every 12 hours on days 1-3. Filgrastim (G-CSF) administered subcutaneously (SC) beginning on day 5 and continuing until blood counts recover then autologous peripheral blood stem cells (PBSC) are harvested, selected for CD34 positive cells, and purged in vitro. If more than 5% of the WBC contains lymphoma cells after induction, then 2 courses of IFF and VP-16 are administered before PBSC harvest.
  Second course: IFF IV continuously on days 1-3, mitoxantrone (DHAD) IV on day 1, and G-CSF SC as in first course.
  Third course: Carmustine IV over 1 hour on day -6, ARA-C and VP-16 IV every 12 hours on days -5 to -2, and melphalan IV on day -1. PBSC are reinfused on day 0. G-CSF is administered SC beginning on day 0 and continuing until blood counts recover. Each course lasts 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Filgrastim (G-CSF); Drug: Carmustine; Drug: Cytarabine (ARA-C); Drug: Etoposide (VP-16); Drug: Ifosfamide; Drug: Melphalan; Drug: mitoxantrone hydrochloride (DHAD); Procedure: Peripheral Blood Stem Cell Transplantation
- Arm II (Experimental): IDSHAP during 4 week courses 2 and 5, MBIDCOS during courses 3 and 6, and IFF and VP-16 IV over 1 hour on days 1-3 and DHAD IV over 15 minutes on day 1 during courses 1, 4, and 7.
  Interventions: Biological: Bleomycin Sulfate (BLM); Biological: Recombinant Interferon Alfa; Drug: Cisplatin (CDDP); Drug: Cyclophosphamide; Drug: Idarubicin; Drug: Leucovorin Calcium; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Vincristine Sulfate; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Bleomycin Sulfate (BLM)
  Other Names: Blenoxane; BLM
  Arms: Arm II
Biological: Filgrastim (G-CSF) — Arm 1: Administered subcutaneously (SC) beginning on day 5 and continuing until blood counts recover through Course 1 then 2 courses administered before PBSC harvest and same regimen with Course 2, then daily with Day 0 of infusion.
  Other Names: G-CSF; Neupogen
  Arms: Arm I
Biological: Recombinant Interferon Alfa
  Arms: Arm II
Drug: Carmustine — Arm 1, Course 3, IV over 1 hour on day -6.
  Other Names: BiCNU; BiCNUI
  Arms: Arm I
Drug: Cisplatin (CDDP)
  Other Names: Platinol; Platinol-AQ
  Arms: Arm II
Drug: Cyclophosphamide
  Other Names: Cytoxan; Neosar
  Arms: Arm II
Drug: Cytarabine (ARA-C) — Arm 1, Course 3, every 12 hours on days -5 to -2.
  Other Names: ARA-C; Cytosar; DepotCyt; Cytosine arabinosine hydrochloride
  Arms: Arm I
Drug: Etoposide (VP-16) — Course 1, IV over 2 hours every 12 hours on days 1-3; Course 3, every 12 hours on days -5 to -2.
  Other Names: VePesid
  Arms: Arm I
Drug: Idarubicin
  Other Names: Idamycin
  Arms: Arm II
Drug: Ifosfamide — During Course 1, IV continuously; Course 2, IV continuously on days 1-3.
  Other Names: Ifex
  Arms: Arm I
Drug: Leucovorin Calcium
  Other Names: Leucovorin; Citrovorum; Wellcovorin
  Arms: Arm II
Drug: Melphalan
  Other Names: Alkeran
  Arms: Arm I
Drug: Methotrexate
  Arms: Arm II
Drug: Methylprednisolone
  Other Names: Depo-Medrol; Medrol; Solu-Medrol
  Arms: Arm II
Drug: mitoxantrone hydrochloride (DHAD) — Arm 1, Course 2, IV on day 1.
  Other Names: mitoxantrone; Novantrone
  Arms: Arm I
Drug: Vincristine Sulfate
  Arms: Arm II
Procedure: Peripheral Blood Stem Cell Transplantation — Infusion of stem cells on Day 0.
  Other Names: autologous peripheral blood stem cells; PBSC
Radiation: Radiation Therapy
  Other Names: RT
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of two regimens of combination chemotherapy in treating patients who have intermediate-grade or immunoblastic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of early intensification vs alternating triple chemotherapy in patients with intermediate-grade or immunoblastic lymphoma with poor prognostic features.
* Compare, in a prospective manner, the cost/benefit ratio of these regimens in these patients.
* Determine the value of monitoring minimal residual disease detection via in vitro culture methods and polymerase chain reaction analysis of peripheral stem cell apheresis products and by longitudinal monitoring of blood and bone marrow samples in these patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are stratified according to tumor score (3 or 4 vs 5 or 6).

During the first course of induction, patients receive IDSHAP comprising idarubicin (IDA) and cisplatin IV continuously on days 1-4, cytarabine (ARA-C) IV over 2 hours on day 5, and methylprednisolone (MePRDL) IV over 15 minutes on days 1-5. During the second course of induction, patients receive MBIDCOS comprising vincristine, bleomycin, and cyclophosphamide IV over 15 minutes on day 1, IDA IV continuously and MePRDL IV over 15 minutes on days 1-3, methotrexate (MTX) IV over 2 hours on day 10, and oral leucovorin calcium every 6 hours on days 11 and 12. Each course lasts 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients with stable or responding disease after induction are randomized to 1 of 2 treatment arms.

Arm I

* Patients receive the following 3 courses of early intensification.

  * First course: Patients receive ifosfamide (IFF) IV continuously and etoposide (VP-16) IV over 2 hours every 12 hours on days 1-3. Filgrastim (G-CSF) is administered subcutaneously (SC) beginning on day 5 and continuing until blood counts recover and then autologous peripheral blood stem cells (PBSC) are harvested, selected for CD34 positive cells, and purged in vitro. If more than 5% of the WBC contains lymphoma cells after induction, then 2 courses of IFF and VP-16 are administered before PBSC harvest.
  * Second course: Patients receive IFF IV continuously on days 1-3, mitoxantrone (DHAD) IV on day 1, and G-CSF SC as in the first course.
  * Third course: Patients receive carmustine IV over 1 hour on day -6, ARA-C and VP-16 IV every 12 hours on days -5 to -2, and melphalan IV on day -1. PBSC are reinfused on day 0. G-CSF is administered SC beginning on day 0 and continuing until blood counts recover. Each course lasts 3 weeks in the absence of disease progression or unacceptable toxicity.

Arm II

* Patients receive IDSHAP during courses 2 and 5, MBIDCOS during courses 3 and 6, and IFF and VP-16 IV over 1 hour on days 1-3 and DHAD IV over 15 minutes on day 1 during courses 1, 4, and 7. Each course lasts 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients with residual disease after completion of arm I or II treatment undergo radiotherapy to areas of bulk disease if feasible. Patients on both arms with meningeal involvement receive ARA-C intrathecally (IT) alternated with MTX every other day until 1 week after clearing of CNS disease and then 2 IT injections during every course of chemotherapy thereafter. Patients with divergent histology who achieve complete response after completion of arm I or II treatment receive interferon alfa 3 times a week for 1 year.

Patients are followed at 1 month, every 3 months for 1 year, every 6 months for 1 year, and then annually for 2 years.

PROJECTED ACCRUAL: A maximum of 136 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of previously untreated intermediate-grade or immunoblastic lymphoma

  * Tumor score of 3 or greater, defined by the presence of 3 or more of the following criteria :

    * Ann Arbor stage III or IV disease
    * B symptoms (fever, sweats, and weight loss greater than 10%)
    * At least 1 tumor mass greater than 7 cm or mediastinal mass visible on plain chest x-ray
    * Beta-2 microglobulin at least 3.0
    * Lactic dehydrogenase at least 1.1 times the upper limit of normal
* T- and B-cell lymphomas allowed if intermediate grade or immunoblastic
* Divergent histologies, including bone marrow involvement, allowed
* CNS involvement allowed NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 15 to 59

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2.0 mg/dL (unless elevation due to lymphoma)

Renal:

* Creatinine no greater than 1.5 mg/dL (unless elevation due to lymphoma)

Cardiovascular:

* LVEF greater than 50% by echocardiogram if over age 45
* No congestive heart failure, angina, history of myocardial infarction, or arrhythmia unless cleared by principal investigator after cardiology consultation

Pulmonary:

* No history of chronic obstructive or restrictive lung disease
* Pulmonary consultation required for smokers or patients with questionable lung function

Other:

* HIV negative
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior malignancy with poor prognosis (less than 90% probability of surviving for 5 years)
* No geographic, economic, emotional, or social condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* No prior endocrine therapy

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 1995-10-30 (Actual); Primary Completion 2004-02-04 (Actual); Study Completion 2004-02-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of Early Intensification vs. Alternating Triple Chemotherapy | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org